CLINICAL TRIAL: NCT03521349
Title: Correlational and Intervention Effects of Egg Consumption on Macular Carotenoids, Cognition, and Achievement During Childhood
Acronym: SHELL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Principal Investigator, Naiman Khan, Naiman Khan, PhD, RD, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SHELL
Record Dates: First submitted 2018-04-28; First posted 2018-05-11 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Diet Habit; Cognitive Control
Keywords: Electroencephalography; Executive Function; Egg; Diet
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg White Snacks (Placebo Comparator): Egg white-based snacks
  Interventions: Other: Egg White Control
- Whole Egg Snacks (Experimental): Whole egg-based snacks
  Interventions: Other: Whole Egg Intervention

INTERVENTIONS:
Other: Whole Egg Intervention — Participants will consume an isocaloric muffin containing important bioactives from whole eggs.
  Arms: Whole Egg Snacks
Other: Egg White Control — Participants will consume an isocaloric muffin containing egg white, lacking important bioactives from whole eggs.
  Arms: Egg White Snacks

SUMMARY:
The aim of this study is to examine the correlational and intervention effects of egg consumption on macular carotenoids, cognition, and achievement during childhood. Initially, this will be done with correlational examination of egg consumption and macular carotenoids. Individuals with low carotenoid status will be invited to participant in a month-long egg-based dietary intervention aimed at improving carotenoid status.

DETAILED DESCRIPTION:
Identification of foods that promote childhood cognitive function has the potential to have a lasting impact on children's long-term cognitive well-being. The nutrient profile in egg yolks, particularly the xanthophyll lutein, may be uniquely suitable for supporting important cognitive processes including attention, memory, and academic achievement. Lutein is the predominant carotenoid in the brain, comprising up to 77% of carotenoids in the brain. Further, lutein is among three xanthophylls that accumulate as macular pigment and protect the eye against photooxidative damage.

Accordingly, this work aims to: 1) assess the correlational relationship between habitual egg consumption, macular pigment optical density (MPOD), neurocognitive function and achievement among 7-12-years-olds; and 2) conduct a 4-week egg intake randomized controlled intervention (7 whole eggs/week vs 7 egg whites/week) to investigate the effects of regular egg consumption on changes in MPOD and behavioral and neuroelectric measures of cognitive control and relational memory, and academic achievement among school-aged children. Male and female children between 7-12 years (n=240) will be recruited. All children will be allowed (i.e., regardless of level of MPOD) to participate to address aim 1. A subsample of participants (n=80 [40 per group]) with lower MPOD (i.e., ≤0.40) will be invited to enroll in a 4-week egg intake randomized controlled trial. Following baseline testing, participants will be randomly assigned to one of two intervention groups (7 whole eggs/week vs 7 egg whites/week) for a 4- week period.

The investigators hypothesize that greater habitual egg consumption will be positively associated with MPOD and attention and memory and neural efficiency, and academic achievement. Further, the investigators anticipate that consuming whole eggs - via a 4-week intervention - will result in greater gains in behavioral and ERP cognitive measures and academic achievement, relative to egg white consumption. Finally, it is expected that cognitive benefits will correlate with change in MPOD, thereby establishing the importance of whole eggs for cognitive function and academic achievement in childhood.

The successful completion of the proposed work is expected to generate new knowledge establishing the importance of regular whole egg consumption, specifically lutein induced changes in macular carotenoids, for improving performance in cognitive processes vital for learning and long-term scholastic success among school-aged children.

ELIGIBILITY:
Inclusion Criteria:

* a. Parental/guardian consent b. Between 7-12 years c. Absence of physician diagnosis of autism spectrum disorder d. Normal or corrected-to-normal vision based on the minimal 20/20 standard f. Intervention Only: Absence of food allergies

Exclusion Criteria:

* a. Parental/guardian non-consent b. Younger than 7 years or older than 12 years c. Physician diagnosis of autism spectrum disorder d. Uncorrected vision f. Intervention Only: Presence of food allergies

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-03-21 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive control | 1 month
  Changes in Cognitive Task Performance between Groups

SECONDARY OUTCOMES:
Macular Pigment Optical Density (MPOD) | 1 month
  Changes in MPOD between Groups

CONTACTS AND LOCATIONS:
Overall Officials: Naiman Khan, PhD, RD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be disseminated by journal articles, thesis or academic papers, conference presentations, and sharing with the funding organization. No subject's identity will be disclosed in any presentation or released without their written permission.

REFERENCES:
- [Derived] Liu R, Edwards CG, Cannavale CN, Flemming IR, Chojnacki MR, Reeser GE, Iwinski SJ, Renzi-Hammond LM, Khan NA. Weight Status and Visceral Adiposity Mediate the Relation between Exclusive Breastfeeding Duration and Skin Carotenoids in Later Childhood. Curr Dev Nutr. 2021 Feb 15;5(3):nzab010. doi: 10.1093/cdn/nzab010. eCollection 2021 Mar. PMID 33758790